CLINICAL TRIAL: NCT00877409
Title: A Monocentric, Single-Blind, Randomized, Placebo-Controlled Study of the Safety and Efficacy of the Topical Drug Acnase Creme in the Treatment of Acne Vulgaris I and II
Brief Title: Safety and Efficacy Study of Acnase Creme in the Treatment of Acne Vulgaris I and II
Acronym: ACNASE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zurita Laboratorio Farmaceutico Ltda. (Industry)
Responsible Party: Zurita Laboratorio Farmaceutico Ltda., Zurita Laboratorio Farmaceutico Ltda.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EAA461-08/v8; EAA461-08/v8
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Acne Vulgaris
Keywords: Acnase; Acne Vulgaris; Safety; Efficacy
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acnase (Active Comparator)
  Interventions: Drug: Benzoyl Peroxide 5% and Sulphur 2%
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle of Acnase

INTERVENTIONS:
Drug: Benzoyl Peroxide 5% and Sulphur 2% — The product will be applied topically forming a thin layer, 1 time a day (at night) throughout the area affected by lesions.
  Other Names: Acnase
  Arms: Acnase
Drug: Vehicle of Acnase — The product will be applied topically forming a thin layer, 1 time a day (at night) throughout the area affected by lesions.
  Other Names: Control; Vehicle; Placebo
  Arms: Vehicle

SUMMARY:
The objective of this study is to establish the safety in use of the topical drug Acnase Creme and its effectiveness in treatment of acne grade I (comedones) and II (comedones, papules, pustules).

DETAILED DESCRIPTION:
The acne is a common dermatosis in dermatological practice, affects more than 80% of the population during the second and third decades of life. It is found worldwide, with no evidence of racial or ethnic differences that influence the susceptibility to its development. However there is influence of genetic factors, hormones, the use of certain drugs that may have previous or aggravate the disease.

It is an inflammatory disease of the follicle polissebáceo, which consists of large sebaceous glands, multiacinares, rudimentary hair follicle and a channel comprising a acro-infundibulum in its upper portion and an infra-infundibulum in the dermal portion.

This is a benign condition, self-limited, but can cause serious psychological problems or disfiguring scars, which can persist for the rest of life.

The initial change is a disorder of follicular epithelial differentiation, during which the cornea cells (keratinocytes) which are the follicle polissebáceo are excessively released in the lumen. The result of this event is the appearance of the precursor, microcomedão, from which the lesions of acne are developed (closed comedones, open comedones, papules, pustules and nodules). The dilation of the follicular infundibulum with the material produces a corneal comedão closed. This is the first clinically visible lesions of acne. As hyperkeratosis extends to the upper infundibulum, extended its opening, it formed the comedão open.

The pathogenesis of acne is complex and understood only in part. The follicular occlusion with adherent keratinocytes and activation of hormone secretion resulting in the formation of sebaceous microcomedão. Studies suggest that free fatty acids intrafoliculares control inflammation through chemotactic properties on leukocytes, monocytes and neutrophils. The free fatty acids may provide the primary stimulus for the retention hyperkeratosis follicularis. Moreover, tallow provides a favorable substrate for the proliferation of Propiniobacterium acnes (P. acnes). Studies suggest that P. acnes, a microaerophilic bacterium (almost anaerobic), Gram-positive, has a lipase able to hydrolyze triglycerides in sebum into free fatty acids. Therefore, these pathogens play critical role in the generation of inflammatory lesions. The P. acnes produces proteases and neuroaminidases, which may increase the permeability of the follicular epithelium. Also produce a chemotactic factor of low molecular weight that selects the polymorphonuclear leukocytes. In the process of phagocytosis of bacteria are released hydrolases, which break the integrity of the follicular wall. Subsequently, the content intrafolicular - fragments of keratin, fat, hair, and P. acnes - is expelled to the dermis.

If surface aggregation of neutrophils, as was a wheal, and with the presence of purulent secretion, a pustule. With the infiltration of inflammation deep and extensive, a nodule or cyst is produced.

Clinically, the eruption acnéica is located predominantly in the face (90%) and to a lesser extent, in the back (60%) and chest (15%). As young man, mainly affects the face, while in older, the back.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12 to 35 years;
* Oily skin with tendency to acne;
* Presence of non-inflammatory lesions and inflammatory, acne vulgaris diagnosed as grade I or II, as the following: I) Comedones - only comedones; II) Papulopustular - comedones, papules and pustules; III) Nodulocystic - comedones, papules, pustules, nodules and cysts; IV) Conglobates - severe acne, usually affects other areas of the body, out of preference, giving comedones, papules, pustules, abscesses, confluent nodules, cysts and scars.
* Agreement in compliance with the procedures of the trial and attend the clinic on certain days and times for medical evaluations and scores of injuries acne;
* Signing of the Term of Free and Informed Consent and agreement of the lowest in the case of patients between 12 and 17 years.

Exclusion Criteria:

* Pregnancy (pregnancy test by urinary indication to women voluntary of childbearing age);
* Nursing;
* Nodulocystic and Conglobates acne;
* Conditions associated hormone (tireoid disease, micropolicysts ovaries, adrenal or pituitary disorders);
* Drug use systemic corticosteroids, anticonvulsants, photo-sensibility and / or new drugs for up to 01 months before the selection;
* Use of topical therapy, systemic or physical (cleaning of the skin) for the treatment of acne at least 01 months before the selection;
* History of atopic or allergic skin;
* History of hypersensitivity to Benzoyl peroxide or sulfur;
* Skin Conditions active (and / or spread) that may interfere with the outcome of the study;
* Beginning or end-use of contraceptives; (for females)
* Sunlight intense exposure until 01 months before the assessment;
* Aesthetic treatments, skin up to 01 months before the selection;
* Use of specific oily cosmetic for skin / acne and makeup, facial moisturizing, etc..;
* Use of the drug Acnase prior to inclusion in the study.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Average clinical development of target lesions of the groups for each experimental time. | 12 weeks

SECONDARY OUTCOMES:
Clinical evolution of the acne through the counting of inflammatory and non - inflammatory lesions. | 12 weeks
Evaluation of oily skin through the clinical evaluation with four-point scale (absent, mild, moderate, intense) | 12 weeks
Observation of occurrence and intensity of clinical parameters erythema, scaling, itching and burning through the clinical evaluation with four-point scale (absent, mild, moderate, severe). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Schalka, MD, Principal Investigator — Medcin Instituto da Pele Ltda
Locations (1):
- Medcin Instituto da Pele Ltda., Osasco, São Paulo, Brazil